CLINICAL TRIAL: NCT06211920
Title: Prehospital Use of Non-invasive Ventilation for Acute Respiratory Failure Due to Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: Prehospital Non-invasive Ventilation for Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Acronym: PRENIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Denmark Region (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 97289
Record Dates: First submitted 2023-12-07; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: COPD Exacerbation; COPD Exacerbation Acute; Noninvasive Ventilation; Emergency Medical Services
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: Investigator-initiated, randomized 1:1, clinical trial
Masking Description: Due to the nature of the intervention, the clinicians performing the intervention cannot be blinded. This is also the case for patients along with any legally designated representatives at the scene. As it is common to note the prehospital treatment in the patient's medical records clinicians at the ED and/or ICU will not necessarily be blinded either. For the same reason, investigators involved in data entry will also not be blinded meaning that outcomes such as change in arterial pH are entered without blinding. However, there is little - if any - subjectivity in evaluating these outcomes and blinding is therefore likely of minor importance.
  A patient - or alternatively the consenting legally designated representatives - will not be informed of the allocation until the end of follow-up and only per request on the consent form.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-invasive ventilation (NIV) + standard medical treatment (Experimental): The intervention will consist of application of NIV through a facemask. This will happen as soon as possible after the patient has been randomized by opening the opaque envelope. All patients will receive the same standardized ventilator settings at initiation. The IPAP will be set at 12 cm H2O and the PEEP at 5 cm H2O. These settings are preset on the ventilator used in the physician manned mobile emergency care unit (MECU) in the Central Denmark Region. Oxygen delivery will be adjusted to an arterial oxygen saturation of 88-92%. Further adjustment of ventilator settings and evaluation of treatment effect will be at the discretion of the prehospital physician.
  NIV will be administered together with standard medical treatment described below.
  Interventions: Other: Non-invasive ventilation
- Standard medical treatment alone (No Intervention): The standard treatment may include inhaled bronchodilators, intravenous corticosteroids, and titrated oxygen supplementation. Although this treatment is based on regional standard operating procedures (SOP), it may differ from patient to patient because it is based on the clinical judgement by the emergency physician in the MECU.
  Inhaled bronchodilators can be given in the form of Fenoterol and Ipratropium as a combination drug and/or Salbutamol. Both as a nebulizer solution. One dose (4 ml) of the combination drug contains 1,25 mg Fenoterol and 0,5 mg Ipratropium. Salbutamol will be administered in a concentration of 1 mg/ml. Five mg will be given initially, which can be repeated if necessary.
  Corticosteroids can be given in the form of Methylprednisolone 40-80 mg administered intravenously after establishing an intravenous access.
  Oxygen therapy will be delivered through a nasal cannula if possible or a non-rebreather mask to maintain an arterial saturation of 88-92%.

INTERVENTIONS:
Other: Non-invasive ventilation — The application of NIV will be performed using af a facemask as soon as possible after the patient has been randomized by opening the opaque envelope. All patients will receive the same standardized ventilator settings at initiation. The IPAP will be set at 12 cm H2O and the PEEP at 5 cm H2O. Oxygen delivery will be adjusted to an arterial oxygen saturation of 88-92%. Further adjustment of ventilator settings and evaluation of treatment effect will be at the discretion of the prehospital physician.
  Other Names: Standard medical treatment alone
  Arms: Non-invasive ventilation (NIV) + standard medical treatment

SUMMARY:
The goal of this clinical trial is to test if treatment with prehospital Non-invasive ventilation (NIV) for patients with acute respiratory failure (ARF), due to acute exacerbation of chronic obstructive pulmonary disease (AECOPD) based on in-hospital criteria, should be used in the prehospital setting. This is performed with the introduction of prehospital arterial blood gas analyzation. The primary objective is:

• To determine if early prehospital applied NIV together with standard medical treatment will affect arterial pH at hospital arrival in patients with ARF due to AECOPD.

Participants in the intervention will receive Non-invasive ventilation together with standard medical treatment. The intervention will be compared to standard medical treatment alone, that may include inhaled bronchodilators, intravenous corticosteroids, and titrated oxygen supplementation.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years.
2. Medical history of COPD.
3. Unable to give informed consent ("Inhabil" in Danish) based on the criteria below
4. Respiratory acidosis with a PaCO2 of > 6,0 kPa and a pH of < 7,30.

   And one of the following:
5. Respiratory rate of > 25 per minute.
6. Hypoxia with a PaO2 < 7 kPa and/or a saturation < 88% without oxygen administered.

Exclusion Criteria:

1. Upper gastrointestinal hemorrhage or vomiting.
2. Anatomical abnormality that precludes the use of an oro-nasal interface.
3. Suspicion of pneumothorax.
4. Cardiac or respiratory arrest.
5. Uncontrollable malignant arrhythmia.
6. Refractory shock (systolic blood pressure < 90 mmHg) despite fluids and/or vasoactive drugs given.
7. Required orotracheal intubation.
8. Suspected upper airway obstruction.
9. No indication for life-prolonging treatment with NIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
The change in pH observed during the prehospital treatment period. | During the prehospital treatment for a maximum of 2 hours.
  pH will be measured before randomization in the prehospital setting and at arrival at the emergency department. The change in pH will be compared between the two groups.

SECONDARY OUTCOMES:
Overall time with a NIV-mask on. | From time of randomization and during the entire admission. Assessed up to 30 days.
  NIV treatment time will be registrered in both groups on a schematic form. The outcome will be compared between the two groups.
Proportion treated with invasive respiratory treatment. | During both the prehospital treatment and the entire hospital admission. Assessed up to 30 days.
  The outcome will be compared between the two groups.
Length of hospital stay. | From time of admission and up until discharge. Assessed up to 30 days.
  The outcome will be compared between the two groups.
The change in pH 2 hours from the initial prehospital ABG analysis. | 2 hours from the initial prehospital ABG analysis.
  pH will be measured before randomization in the prehospital setting and again after 2 hours. The change in pH will be compared between the two groups.
Mortality (in-hospital and 30 days after admission). | During the length of hospital stay and up until 30 days after admission.
  The outcome will be compared between the two groups.
Prehospital treatment time (both on-scene time and transport time). | During the prehospital treatment for a maximum of 2 hours.
  The outcome will be compared between the two groups.

OTHER OUTCOMES:
Correlation between venous and arterial pH. | During the prehospital treatment for a maximum of 2 hours.
Correlation between PaCO2 and the partial pressure of CO2 in venous blood (PvCO2). | During the prehospital treatment for a maximum of 2 hours.
Correlation between "venous to arterial conversion" (v-TAC) and the results from the actual arterial blood gas analysis regarding pH, PaCO2 and PaO2 in all enrolled patients. | During the prehospital treatment for a maximum of 2 hours.
  We will use a mathematical model (v-TAC) to arterialize the results from all the venous blood gas analysis from each enrolled patient. We will correlate these results regarding pH, PaCO2 and PaO2 with the results from the actual ABG analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jesper H Haunstrup Brendel, MD, Principal Investigator — Research and development, The Prehospital Department in The Central Denmark Region
Locations (1):
- Prehospital Emegency Medical Service, Central Denmark Region, Denmark, Aarhus N, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Six months after the publication of the last results, all de-identified individual patient data will be made available for data sharing. Procedures, including re-coding of key variables, will be put in place to allow for complete de-identification of the data. Data will be completely anonymized according to Danish law.
  All relevant trial-related documents, including the protocol, data dictionary, and the main statistical code, will be shared along with the data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: There will be no predetermined end date for the data sharing.
Access Criteria: Data will be available for any research purpose to all interested parties who have approval from an independent review committee and who have a methodological sound proposal as determined by the steering committee of the current trial. Only the methodological qualities and not the purpose or objective of the proposal will be considered. Interested parties will be able to request the data by contacting the principal investigator. Authorship of publications emerging from the shared data will follow standard authorship guidelines from the International Committee of Medical Journal Editors and might or might not include authors from the steering committee depending on the nature of their involvement.